CLINICAL TRIAL: NCT05822557
Title: A Study Evaluating a Newly Designed Nutritional Tube Feeding Pouch for Bolus Feeding in Adults
Brief Title: Bolus Pouch Feed Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BOPFS2020
Record Dates: First submitted 2022-04-12; First posted 2023-04-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cancer; Neurological Disorder; Gastrointestinal Dysfunction; Oral Complication; Stroke
MeSH Terms: conditions — Neoplasms; Nervous System Diseases; Stroke

STUDY DESIGN:
Intervention Model Description: This is a prospective, longitudinal, 28-day intervention study with a 7-day baseline period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bolus Pouch Feed (Experimental): A 250 ml feeding pouch containing 400 kcal.
  Interventions: Other: Bolus Pouch Feed

INTERVENTIONS:
Other: Bolus Pouch Feed — Following the 7-day baseline period, all patients will enter the 28-day intervention period, where they will receive the intervention feed daily. The feed prescription will be determined on an individual basis by the Dietitian responsible for the patient's nutritional management

SUMMARY:
The primary aim of this study is to evaluate the impact of introducing a new enteral tube feed on health and feeding related quality of life. Secondary aims are to assess ease of use, liking, compliance, gastrointestinal tolerance, nutrient intake, anthropometric changes and safety.

DETAILED DESCRIPTION:
Bolus enteral tube feeding (termed 'bolus feeding') is an increasingly common method of providing nutritional support to home enterally tube fed (HETF) patients, particularly those who are more active and/or require greater flexibility in their feeding regimen. However, current methods of bolus feeding are complex to administer, messy, may be unhygienic, and require and lead to a significant amount of plastic waste. Therefore, there is a clear need for a simpler and optimised way to provide bolus feeds. The aim of this study is to evaluate the impact of introducing a new enteral tube feed on health and feeding related quality of life, ease of use, liking, compliance, gastrointestinal tolerance, nutritional intake, anthropometry and safety. This is a prospective, longitudinal, 28-day intervention study with a 7-day baseline period.

ELIGIBILITY:
Inclusion Criteria:

* ≥16 years of age
* Using or requiring an enteral tube feed as part of nutritional management plan
* Using or about to use bolus tube feeding methods at least once daily
* Expected to receive at least 400 kcal/day from the intervention feed
* Written or electronic informed consent from patient, or verbally given consent countersigned by a witness for those physically unable to sign.

Exclusion Criteria:

* Parenteral nutrition contributing more than 70% of total energy requirements
* Patients with major hepatic dysfunction (i.e., decompensated liver disease)
* Patients with major renal dysfunction [i.e., requiring filtration or stage 4/5 chronic kidney disease (CKD)]
* Patients receiving inpatient care
* Participation in other clinical intervention studies within 2 weeks of this study
* Adults lacking mental capacity to consent
* Allergy to any study product ingredients
* Investigator concern regarding ability or willingness of patient to comply with the study requirements.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Health and feeding related quality of life | Baseline to end of intervention (Day 35)
  At baseline, and at the mid-point and end of the intervention period, health and feeding related quality of life will be assessed by the FACT-EQ questionnaire.

SECONDARY OUTCOMES:
Ease of administration | Baseline to end of intervention (Day 35)
  At baseline, and at the mid-point and end of the intervention period, patients and dietitians will be asked to rate the ease of administering the enteral tube feed via a Likert-style questionnaire. Patients will also count the amount of feeding equipment required to administer the enteral feed at baseline, and at the midpoint and end of the intervention period.
Liking of feeding method | Baseline to end of intervention (Day 35)
  At baseline, and at the mid-point and end of the intervention period, patients will be asked to rate their liking of their usual feeding method or of the intervention feed, respectively via a 7-point Likert scale questionnaire.
Gastrointestinal tolerance | Baseline to end of intervention (Day 35)
  A standardised gastrointestinal (GI) tolerance questionnaire to capture perceived severity (none, mild, moderate or severe) of common gastrointestinal symptoms (diarrhoea, constipation, bloating, abdominal discomfort, vomiting and nausea) will be recorded at the end of each week. Information about bowel movements will also be collected using the Bristol Stool Chart©.
Compliance | Baseline to end of intervention (Day 35)
  Compliance with feed prescription will be assessed daily throughout the study by recording how much feed was received, to be recorded by the patient.
Nutrient intake | Baseline to end of intervention (Day 35)
  At baseline, and at the mid-point and end of the intervention period, the dietitian will conduct a 24-h dietary recall with the patient to record all food, drink and nutritional feeds provided in the 24 h prior. Trained research staff will subsequently analyse all records utilising a nutritional software package (Nutritics Professional v3.09, Nutritics, Ireland) for macro- and micro-nutrient intakes.
Body weight (kg) | Baseline to end of intervention (Day 35)
  At baseline and at the end of the intervention period, body weight (kg) will be measured using standard methods to the nearest 0.1 kg using a weighing scale without heavy clothing.
Adverse Events | Baseline to end of intervention (Day 35)
  All adverse events will be recorded throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, PhD, Study Chair — Nutricia UK Ltd
Locations (15):
- United Kingdom (15):
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - County Durham and Darlington NHS Foundation Trust, Darlington
  - NHS Tayside, Dundee
  - Royal Surrey NHS Foundation Trust, Guildford
  - Betsi Cadwaladr University Health Board, Holywell
  - Calderdale & Huddersfield NHS Foundation Trust, Huddersfield
  - Leicestershire Partnership NHS Trust, Leicester
  - North East London NHS Foundation Trust, London
  - Northumbria Healthcare NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Southern Health NHS Foundation Trust, Southampton
  - South Warwickshire NHS Foundation Trust, Warwick

IPD SHARING:
Plan to Share IPD: No